CLINICAL TRIAL: NCT01633255
Title: A Pilot, Open-label, Proof-of-Concept Study of the Use of [18F] Fluciclatide PET/CT Imaging in the Evaluation of Anti-AngiogenicTherapy in Renal Cancers
Brief Title: [18]F-Fluciclatide for Kidney Cancer Imaging Studies and Treatment
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 120120; 12-C-0120
Record Dates: First submitted 2012-06-30; First posted 2012-07-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-04-23

CONDITIONS: Kidney Neoplasms
Keywords: Anti-Angiogenic; Dynamic Contrast Enhanced Magnetic Resonance Imaging; PET/CT Imaging Studies
MeSH Terms: conditions — Kidney Neoplasms | interventions — AH 111585

INTERVENTIONS:
Drug: 18F-Fluciclatide

SUMMARY:
Background:

- The experimental contrast agent [18]F-Fluciclatide is being tested for cancer treatment imaging studies. It is designed to show tumors in which new blood vessels are growing. Imaging studies with [18]F-Fluciclatide may help predict how well a tumor will respond to therapy that will prevent the growth of new blood vessels. Researchers will test [18]F-Fluciclatide before beginning treatment and after the first treatment cycle. Participants may also have a third scan with [18]F-Fluciclatide between 2 and 7 days after starting treatment to look for changes in blood vessel growth early after starting therapy.

Objectives:

- To test the safety and effectiveness of [18]F-Fluciclatide in predicting cancer treatment outcomes.

Eligibility:

- Individuals at least 18 years of age who will have kidney cancer treatment to stop tumor blood vessel growth.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Tumor imaging studies and biopsies will be performed before starting the study.
* Participants will have two positron emission tomography (PET) and computed tomography (CT) scans. [18]F-Fluciclatide will be used for each scan. One scan will happen before the start of cancer treatment, and the second will happen after the first treatment cycle.
* Participants may also have an optional third PET/CT scan with [18]F-Fluciclatide. This scan will take place 2 to 7 days after beginning therapy.
* Depending on the location of the tumor, some participants may have an optional magnetic resonance imaging scan to look for changes in tumor blood flow and size. These scans will be done within 3 weeks of each [18]F-Fluciclatide PET/CT scan.
* The scans will be monitored with regular blood tests and vital signs.
* Participants will be followed for up to 1 year after the study to look for overall disease response to therapy.

DETAILED DESCRIPTION:
BACKGROUND:

* Fluciclatide is a small cyclic peptide containing the RGD tri-peptide, which preferentially binds with high affinity to Alpha(v)Beta(3) integrins, which are up-regulated in and may regulate angiogenesis.
* Alpha(v)Beta(3) integrins are also expressed on certain types of tumor cells, such as renal cell cancer.
* [18F] Fluciclatide (previously known as 18F-AH111585) is a new radiopharmaceutical developed for PET imaging, which targets Alpha(v)Beta(3) receptors.
* Initial and ongoing clinical studies performed in Europe and an ongoing multicenter phase 2 proof-of-concept study (which is currently open at the NIH Clinical Center); demonstrate to date that [18F] Fluciclatide is safe and well tolerated.

PRIMARY OBJECTIVE:

- To determine tumor uptake and retention of [18F] Fluciclatide before and after 1 cycle of treatment with targeted anti-angiogenic therapy in renal cell cancer.

ELIGIBILITY:

* Adult subjects (greater than or equal to18 years old), with documented renal or metastatic renal cancer, with at least one tumor greater than or equal to1 cm in diameter outside of the liver, who are scheduled to enroll in a therapy protocol using an anti-angiogenic agent.
* The subject has a platelet count of >100,000 times 10(6)/L, hemoglobin value of >9 g/dL, prothrombin time (PT) and an activated partial thromboplastin time (aPTT) within <2 times normal limits.
* The subject has not received any targeted anti-angiogenic agents within 60 days prior to pre-treatment (baseline) [18F] Fluciclatide PET imaging.

DESIGN:

This will be a pilot, open-label, proof-of-concept study to assess the magnitude of changes in [18F] Fluciclatide PET tumor uptake following treatment with an anti-angiogenic therapy. We expect to enroll 30 evaluable patients in this single center study. When possible, the data analysis will be stratified based on the anti-angiogenic agent received. Subjects will undergo at least two [18F] Fluciclatide PET/CT imaging studies, one pre-therapy and one following completion of 1 cycle of therapy. An optional early post-therapy (2-7 days post therapy commencement) [18F] Fluciclatide PET/CT may be performed. The magnitude of [18F] Fluciclatide uptake on the preand post- treatment PET/CT studies will be evaluated to determine if there is a measureable difference in uptake. Subjects may also undergo standard of care imaging studies as part of routine tumor assessments specified in referring protocols (e.g. diagnostic CT, FDG-PET/CT, etc). Data from the subject s referring therapy protocol will be reviewed for up to one year after anti-angiogenic therapy initiation to assess for tumor response or progression and its relationship to [18F] Fluciclatide PET/CT imaging. Some patients will also undergo optional DCE-MRI scans of the target lesion and in those subjects a comparison between MR parameters and [18F]

Fluciclatide parameters will be made.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult subjects (greater than or equal to18 years old), with documented renal malignancy or metastatic renal cancer, with at least one tumor greater than or equal to1 cm in diameter (not within the liver), who are scheduled for treatment using an anti-angiogenic therapy agent
* Platelet count of >100,000 times 10(6)/L, hemoglobin value of >9 g/dL, PT and an aPTT < 2 times normal limits.
* Clinically acceptable medical history, physical examination and vital signs findings during the screening period (from <4 weeks before administration of [18F] Fluciclatide); i.e. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
* The subject has had no open surgical wounds in close proximity to the target lesion(s) within 10 days prior to study entry.
* The subject has not had a needle/core biopsy of the target lesion within 10 days of PET/CT imaging.
* The subject has not had radiation therapy to the region of the target lesion.

EXCLUSION CRITERIA:

* The subject is pregnant or nursing.
* The subject is being treated with doses of heparin or warfarin resulting in elevation of PT or aPTT >2 times normal.
* The subject has received any anti-angiogenic agent (e.g. bevacizumab, sorafenib, sunitinib) within 60 days prior to pre-treatment (baseline) [18F] Fluciclatide PE imaging. This stipulation does not apply after the baseline [18F] Fluciclatide PET imaging.
* The subject has any contraindication to any of the study procedures, products used or its constituents (e.g. severe claustrophobia unrelieved by oral anxiolytics).
* The subject is unable to lie still for 75 minutes.

2.1.2.6 The subject is known to have a history of hyper- or hypo-coagulation syndromes resulting in prolongation of bleeding parameters. Such coagulopathies include but are not limited to Von Willebrand disease, Protein C deficiency, Protein S deficiency, Hemophilia A/B/C, Factor-V Leiden, and Bernard-Soulier syndrome.

* The subject has undergone a surgical procedure to the target lesion within 28 days prior to baseline [18F] Fluciclatide administration OR is scheduled to undergo a surgical procedure between the baseline and post 1-cycle [18F] Fluciclatide PET/CT.
* The subject has only bone metastasis

ADDITIONAL EXCLUSION CRITERIA FOR SUBJECTS UNDERGOING OPTIONAL MR:

* Serum creatinine within 2 weeks prior to MRI greater than or equal to1.8mg/dl OR estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m(2).
* The subject has known allergy to gadolinium

2.1.3.3 The subject has contraindications to MRI

* Subjects must weigh <136 kg (weight limit for scanner table).
* Subjects cannot have pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04-18; Primary Completion 2014-04-23 (Actual); Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
To determine tumor uptake and retention of [18F] Fluciclatide before and after 1 cycle of treatment with targeted anti-angiogenic therapy in renal cell cancer.

SECONDARY OUTCOMES:
Safety of multiple IV admin. of agent.
Compare data on agent as a PD marker and SOC imaging markers of CR.
Compare DCEMRI parameters with agent PET uptake and retention.
Compare uptake and retention of agent at baseline and at the end of cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Liza Lindenberg, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Egeblad M, Werb Z. New functions for the matrix metalloproteinases in cancer progression. Nat Rev Cancer. 2002 Mar;2(3):161-74. doi: 10.1038/nrc745. PMID 11990853
- [Background] Brooks PC, Clark RA, Cheresh DA. Requirement of vascular integrin alpha v beta 3 for angiogenesis. Science. 1994 Apr 22;264(5158):569-71. doi: 10.1126/science.7512751.
- [Background] Line BR, Mitra A, Nan A, Ghandehari H. Targeting tumor angiogenesis: comparison of peptide and polymer-peptide conjugates. J Nucl Med. 2005 Sep;46(9):1552-60. PMID 16157540